CLINICAL TRIAL: NCT00382421
Title: Swiss Interventional Study on Silent Ischemia (SWISSI 1)
Brief Title: Study to Investigate Effects of Antiischemic Drug Therapy in Silent Ischemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2006-09-28; First posted 2006-09-29 (Estimated); Last update posted 2006-10-12 (Estimated); Status verified 2006-10

CONDITIONS: Myocardial Ischemia
Keywords: Myocardial Ischemia; Randomized Controlled Trials; Drug Therapy
MeSH Terms: conditions — Myocardial Ischemia | interventions — Bisoprolol; Amlodipine; Molsidomine; Aspirin

INTERVENTIONS:
Drug: bisoprolol
Drug: amlodipine
Drug: molsidomine
Drug: acetylsalicylic acid

SUMMARY:
There is a lack of data on the prognostic importance of silent ischemia in totally asymptomatic subjects without history of coronary artery disease (CAD), and, particularly, on a possible benefit of medical therapy in such patients. SWISSI 1 therefore recruits totally asymptomatic subjects older than 40 years of age without any history of CAD but one cardiovascular risk factor with documented silent ischemia. Participants are randomized to open antianginal drug therapy and risk factor control versus only risk factor management and followed up for ≥ 10 years.

DETAILED DESCRIPTION:
Although there is still controversy regarding why ischemic episodes are symptomatic in some patients and completely asymptomatic in others, it is now widely accepted that silent ischemia, like symptomatic episodes, negatively affects prognosis. Silent ischemia may occur in totally asymptomatic patients without (type I) or with a history (type II) of an ischemic cardiac event and coexists with symptomatic episodes in many patients (type III). However, there is a lack of data on the prognostic importance of silent ischemia in totally asymptomatic subjects without history of coronary artery disease (CAD), i.e. silent ischemia type I, and, particularly, on a possible benefit of medical therapy in such patients. Reasons lie in the difficulty to identify such patients and their expected low event rates implying that large patient populations and/or long follow-up periods would be necessary to come to definite conclusions. Still, to address this problem, we perform SWISSI 1 which includes totally asymptomatic subjects older than 40 years of age without any history of CAD but one cardiovascular risk factor with documented silent ischemia. They are randomized to open antianginal drug therapy and risk factor control versus only risk factor management and followed up for ≥ 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented silent myocardial ischemia type I
* At least one cardiovascular risk factor

Exclusion Criteria:

* History of cardiovascular disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1992-02; Study Completion 2006-04

PRIMARY OUTCOMES:
Combination of cardiac death, non-fatal myocardial infarction, unstable angina pectoris, and revascularization

SECONDARY OUTCOMES:
Overall mortality
Cardiac death
Non-fatal myocardial infarction
Stable and unstable angina pectoris
Revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Paul Erne, MD, Principal Investigator — Department of Cardiology, Hospital Lucerne; Paul Erne, MD, Study Chair — Department of Cardiology, Hospital Lucerne
Locations (1):
- Department of Cardiology, Hospital Lucerne, Lucerne, Canton of Lucerne, Switzerland

REFERENCES:
- [Derived] Schoenenberger AW, Jamshidi P, Zuber M, Stuck AE, Pfisterer M, Erne P. Coronary artery disease is common in asymptomatic patients with signs of myocardial ischemia. Eur J Intern Med. 2009 Oct;20(6):607-10. doi: 10.1016/j.ejim.2009.04.001. Epub 2009 May 8. PMID 19782922